CLINICAL TRIAL: NCT04705467
Title: A Multi-Modality Comparison of Needle Placement During Gynecological Brachytherapy Procedures
Brief Title: 3DUS Imaging of Needles in Gynecological Brachytherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 10812
Record Dates: First submitted 2020-12-16; First posted 2021-01-12 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2024-11

CONDITIONS: Gynecologic Cancer
Keywords: 3D Ultrasound; Intervention

STUDY DESIGN:
Intervention Model Description: Patients who are assigned to gynecological brachytherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Other): Device: Gynecological brachytherapy requiring an Interstitial or ring and tandem insert involves insertion of the needle and applicators with no standard real-time image guidance. Occasionally 2-dimensional ultrasound is used, but it greatly limited by its flat nature, preventing a volumetric view of the needle pathways. Interstitial brachytherapy is done under general anesthesia. The trans-abdominal and trans-rectal standard 2D ultrasound that are used in some cases, will be expanded to 3D dimensional imaging through the use of an investigational device. Pre-procedure imaging in the form of MRI is used to help guide needles insertion as well as the clinical exam. Post-procedure CT is done for radiation planning.
  Interventions: Device: Gynecological brachytherapy

INTERVENTIONS:
Device: Gynecological brachytherapy — Management of gynecological malignancies is done through brachytherapy treatment, which involves the delivery of radiation via radioactive sources that are placed into or in close proximity to the tumour.

SUMMARY:
Brachytherapy treatment in gynecological cancers is an essential component to delivering adequate doses of radiation to a tumour while sparing normal tissue. Interstitial or intra-cavitary brachytherapy are often needed in advanced or recurrent disease, in cases where intrauterine brachytherapy may not deliver the optimal outcome. Interstitial or intra-cavitary brachytherapy are based on a defined template-and-needle system, and the procedure relies on clinical examination and pre-treatment imaging to guide needle insertion. There is currently no standard image-guided process to help direct needles in the pelvis. We propose using 3D ultrasound to provide real-time imaging for the brachytherapy procedure, which will aid in avoiding needle insertion into pelvic organs and result in optimal dose coverage to the tumour.

ELIGIBILITY:
Inclusion Criteria:

* Females of age eighteen (18) or greater.
* Patients with locally advanced or recurrent gynecological malignancies who are offered interstitial or ring and tandem brachytherapy treatment. These typically would include patients with primary or recurrent vaginal cancers, endometrial cancers or cervical cancers. Histologies of these cancers are typically adenocarcinomas or squamous cell carcinomas

Exclusion Criteria:

• Above patients who are not offered interstitial brachytherapy as a treatment modality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Needle Localization Accuracy | 16 Months
  Observed needle locations in 3-D TVUS and CT planning images are measured and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- London Regional Cancer Program, Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No